CLINICAL TRIAL: NCT06439758
Title: Effects of First-Line Oral Hypoglycemics in Bone Markers of Treatment Naïve Saudi Adults With Type 2 Diabetes
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Mohammed Ali Almosfer, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB log Number: 2024-6
Record Dates: First submitted 2024-05-20; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Type 2; Osteoporosis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Osteoporosis | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin (Experimental): Metformin is an antihyperglycemic agent which improves glucose tolerance in patients with type 2 diabetes, lowering both basal and postprandial plasma glucose.
  Interventions: Drug: Metformin
- Lifestyle (Placebo Comparator): The effect is when a person's physical or mental health appears to improve after changing their diary system.
  Interventions: Behavioral: Lifestyle

INTERVENTIONS:
Drug: Metformin — Metformin 1000 mg/day for 6 months
  Arms: Metformin
Behavioral: Lifestyle — Dietary lifestyle modifications
  Arms: Lifestyle

SUMMARY:
Both diabetes mellitus and osteoporosis are prevalent diseases with crucial associated mortality and morbidity. There is no clear relevance between bone diseases and diabetes mellitus. Previous research indicates that diabetes and complications related to this disease can contribute to bone disease and DM can also determine bone health. Both kinds of diabetes mellitus bring fracture risk, the most substantial clinical osteoporosis endpoint, which has crucial impact on mortality and morbidity including quality of life of an individual. Although research shows that there is association between Type 1 diabetes (T1DM) and decreased bone mineral density (BMD) values, patients with Type 2 diabetes (T2DM) have either normal or higher than expected BMD values usually. General Objective: To determine the influence of first-line anti-DM therapies in bone turnover markers and metabolism among T2DM naïve Saudi adults.

Specific objectives:

* To investigate the differences in the 3- and 6-month effects of metformin alone, lifestyle intervention alone and combination (metformin + lifestyle modification) on bone markers in T2DM naïve Saudi adults.
* To investigate the differences in the 3- and 6-month effects of metformin alone, lifestyle intervention alone and combination (metformin + lifestyle modification) on metabolism in T2DM naïve Saudi adults.

DETAILED DESCRIPTION:
Design and Setting The present investigation is a multi-center intervention study to be conducted in Hail, Saudi Arabia. The primary endpoint of the study is changes in bone markers.

Participants

Consenting Saudi adults, males, and females, aged 25-65 years with newly diagnosed T2DM will be included. T2DM diagnosis will be done by collaborating primary care physicians following the American Diabetes Association (ADA) and World Health Organization (WHO) criteria:

Fasting plasma glucose ≥7.0mmol/l or ≥126mg/dl. Fasting is defined as no caloric intake for at least 8 hours OR

• 2-h PG ≥200 mg/dl (11.1 mmol/L) during OGTT. The test should be performed as described by WHO, using a glucose load containing the equivalent of 75g anhydrous glucose dissolved in water.

OR • Hba1c ≥6.5% (48 mmol/mol). The test should be performed in a laboratory using a method that is National Glycohemoglobin Standardization Program (NGSP) certified and standardized to the Diabetes Control and Complications (Trial) DCCT assay.

OR

• In a patient with classic symptoms of hyperglycemia or hyperglycemic crisis, a random plasma glucose ≥200 mg/dl (11.1 mmol/L).

Exclusion Criteria

* Non-Saudis and those outside the age range (less than 25 years and above 65 years old).
* Those with comorbidities and existing complications (osteoporosis, uncontrolled hypertension, atherosclerosis, renal and liver abnormalities, morbidly obese, psychologically incapacitated).
* Known cases of T2DM who are already on medications.
* Participants who will be unable to commit to the treatment allocated for 6 months, either for personal reasons or physician's advice.

Intervention

Participants will be assigned to receive, for 6 months either A) Metformin 500mg/day, B) Lifestyle Modification or C) Metformin + Lifestyle Modification. The lifestyle modification management was based on a T2DM prevention program for people with prediabetes and includes weight reduction to 5% from baseline, moderate exercise (150min/week), reduction of fat intake and increased fiber intake (15g/1000kcal). Monitoring will be done at baseline, after 3 months and after 6 months. Below is the schematic diagram of the study:

Figure 1: Schematic diagram of the intervention study.

Data Collection A generalized questionnaire will be administered to patients at baseline which includes demographics, medical history and risk for osteoporosis.

Anthropometrics Height (cm) and weight (kg) will be measured with the participant wearing light clothing. Waist (cm) and hip (cm) circumferences will be measured using standard tape measure. Blood pressure (mmHg) will be measured using a digital sphygmomanometer twice at 15min interval and the average will be recorded.

Sample Collection Fasting blood samples will be collected from participants at baseline and follow-up visits. Routine blood tests (Glucose/HbA1c, liver function tests, renal function tests, and lipid profile) will be done at primary healthcare will be measured using the ARCHITECT c4000 clinical chemistry analyzer and Abbott Afinion HbA1c analyzer. For the bone markers (CTX, PINP, Sclerostin, and Osteocalcin) will be sent to the Chair for Biomarkers of Chronic Diseases (CBCD) in King Saud University, Riyadh, Saudi Arabia for testing using the enzyme-linked immunosorbent assay (ELISA). CTX and PINP will be measured using Cobas e411 immunoassay analyzer. Sclerostin, and Osteocalcin (NMID)will be measured using commercially available assays.

Sample size calculation Mori et al. (2017) have reported the significant decrease in CTX after 3-months in participants consuming metformin as compared to participants consuming pioglitazone with the effect size of 0.40. In our study, to determine the significant change in BTM with the effect size of 0.30 with the power of 80% the required total sample size would be 111 at 95% CI divided in 3 groups (N=37 per group). We intend to recruit 40 participants or more per group to account for dropouts.

Data Analysis Data analysis will be done using SPSS (version 21, Chicago, IL, USA). Statistical analysis will be performed using Intent-to-Treat analysis. All normally distributed data will be presented as mean and standard deviations, while non-normally distributed data will be presented as median and interquartile range. Categorical data will be presented as frequencies and percentages (%). Analysis of Variance (ANOVA) and Kruskal Wallis tests will be used to compare significant baseline differences between groups. Log transformation will be used to transform non-normal variables prior to repeated measure analysis of variance ANOVA, which will be used to obtain within group differences. Logistic regression analysis showing odds of improvement in bone markers as well as other variables of interest in groups will be calculated. A p-value <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Consenting Saudi adults, males, and females, aged 25-65 years with newly diagnosed T2DM will be included.
* T2DM diagnosis will be done by collaborating primary care physicians following the American Diabetes Association (ADA) and World Health Organization (WHO) criteria (ADA, 2022):
* Fasting plasma glucose ≥7.0mmol/l or ≥126mg/dl. Fasting is defined as no caloric intake for at least 8 hours OR
* 2-h PG ≥200 mg/dl (11.1 mmol/L) during OGTT. The test should be performed as described by WHO, using a glucose load containing the equivalent of 75g anhydrous glucose dissolved in water.

OR •Hba1c ≥6.5% (48 mmol/mol). The test should be performed in a laboratory using a method that is National Glycohemoglobin Standardization Program (NGSP) certified and standardized to the Diabetes Control and Complications (Trial) DCCT assay.

OR

•In a patient with classic symptoms of hyperglycemia or hyperglycemic crisis, a random plasma glucose ≥200 mg/dl (11.1 mmol/L).

Exclusion Criteria:

* Non-Saudis and those outside the age range (less than 25 years and above 65 years old).
* Those with comorbidities and existing complications (osteoporosis, uncontrolled hypertension, atherosclerosis, renal and liver abnormalities, morbidly obese, psychologically incapacitated).
* Known cases of T2DM who are already on medications.
* Participants who will be unable to commit to the treatment allocated for 6 months, either for personal reasons or physician's advice.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes in bone marker CTX post intervention | 6 months
  Changes in CTX (pg/mL)
Changes in bone marker PINP post intervention | 6 months
  Changes in PINP (ug/L)
Changes in bone marker Sclerostin post intervention | 6 months
  Changes in Sclerostin (pmol/L)
Changes in bone marker Osteocalcin post intervention | 6 months
  Changes in Osteocalcin (ng/mL)

SECONDARY OUTCOMES:
Changes in fasting glucose, urea, and lipid profile post intervention | 6 months
  changes in Lipid profile (HDL, total cholesterol, Triglycerides), Urea, and fasting Glucose (all mmol/L)
Changes in Creatinine post intervention | 6 months
  Changes in Creatinine (umol/L)
Changes in Liver profile post intervention | 6 months
  Changes in AST, and ALT (U/L)

CONTACTS AND LOCATIONS:
Overall Officials: Nassir Mo Al-dagari, PhD, Study Director — King Saud

IPD SHARING:
Plan to Share IPD: No